CLINICAL TRIAL: NCT06447948
Title: Keep Exercising & Stay Steady (KESS): Development and Feasibility of a Digital Health Intervention to Encourage Exercise Maintenance After Fall Prevention Exercise Programmes End
Brief Title: Keep Exercising & Stay Steady: Development and Feasibility of a Digital Health Intervention to Encourage Exercise Maintenance After Fall Prevention Exercise Programmes End.
Acronym: KESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Orthopaedic Research UK (Unknown); HealthWorks Newcastle Upon Tyne (Unknown); KOKU Health CIC (Unknown); The University of Manchester (Unknown); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Audsley 2024-6365-5990
Record Dates: First submitted 2024-05-13; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Fall Patients
Keywords: Falls Prevention; Ageing Health; Physical activity; Exercise Maintenance; Behaviour Change; Digital health; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Phase 1- Acceptability Study & Phase 2-Feasibility Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Phase 1 (Acceptability Study) intervention arm. Phase 1 participants (n=10) will test the digital health / falls prevention exercise intervention components (e.g. PA via wearables, digital peer support and home exercise delivered via KOKU App) for 1 month.
  Phase 2 (Feasibility Study). Intervention Arm. Phase 2 participants (n=30) will test the optimised digital health / falls prevention exercise intervention components for 6 months.
  Interventions: Behavioral: Keep Exercising and Stay Steady

INTERVENTIONS:
Behavioral: Keep Exercising and Stay Steady — Digital Health, home exercise intervention containing a digital NHS approved falls prevention exercise App (Keep On Keep Up), fitness watches, telephone and/or social media communication, and behavior change techniques.
  Currently (date, 13 May 2024) the intervention has not been developed with the community of practice group. Further details of the phase 1 and phase 2 interventions will be provided after the community of practice events.
  Other Names: KESS

SUMMARY:
Falls and broken bones are a common health problem faced by older adults. Worldwide, one third of adults aged over 65 years old, and half of adults aged over 80 years, fall each year. One in five falls in older adults result in hospitalisation and one in twenty cause broken bones. Each year, 300,000 older adults break a bone following a fall which costs the UK £4.4billion in healthcare costs. Broken hip bones are the most serious outcome of a fall. One in twenty older adults will die and one in five need care assisted living following a hip fracture.

Muscles and bones become weaker after 50 years of age which increases an older adults' risk of falling and breaking a bone. Falls prevention programmes that include muscle strength and balance exercise improves physical function and helps to prevent falls and broken bones in older adults. However, many older adults stop doing exercise and become less physically active after falls prevention programmes end. Gains in balance and muscle strength are lost and falls risk increase if people don't keep exercising. More people are reaching older ages and becoming less active. Therefore, this problem will worsen unless healthcare practices become better at preventing falls and broken bones in older adults.

The research ambition is to create a technology supported home exercise programme that encourages older adults to keep exercising after falls prevention programmes end. This will help to prevent future falls and broken bones which will allow more older adults to continue living independently. The home exercise programme will benefit older adults everyday lives by helping them to maintain good physical health and improve their ability to perform daily tasks without the fear of falling.

Older people at risk of falls, clinicians, and public members will be invited to form a research advisory group. The group will work with the research team to create the home exercise programme and research plan and advise how best to communicate the research to the public. Diversity within the research advisory group will be important to help shape the research to meet the diverse views and needs of the many different people affected by falls and broken bones. We will target the research to help older adults with the greatest health needs. Older adults living in deprived neighbourhoods have the greatest risk of falling and dying following a broken bone. The home exercise programme will be researched in older adults attending falls prevention programmes in the most deprived regions of England. This will help us to explore whether the programme could encourage the continuation of exercise in older adults who need it most.

DETAILED DESCRIPTION:
PURPOSE:

Age-related declines in muscle strength and balance are key risk factors for falls and severe injury in older adults. Completion of group-based Falls Management Exercise (FaME) programmes, significantly improves muscle strength and balance, functional status and reduces falls incidence and injurious falls in older adults. Significant reductions in falls incidence are sustained for up to 2 years in people who maintain increases in their physical activity (PA) levels after FaME programmes end (IRR=0.49, 95% CI 0.30, 0.79; p=0.004). The proportion of people considered as being physically active is 54% upon exiting FaME programmes. However, these proportions decrease to between 40% to 49%, six to eighteen months after FaME programmes end.

Over time, improvements in strength, balance and physical function are lost and falls incidence increase if people do not remain active after programmes end. Home-based exercise delivered via digital means is effective at improving strength, balance and functional status and significantly reduces falls incidence in older adults. This research aims is to develop and investigate the feasibility and acceptability of a digitally supported exercise maintenance intervention, that includes an NHS Approved Falls Prevention App (Keep on Keep Up (KOKU) App) and PA monitoring tools, to people exiting FaME programmes.

STUDY AIM: To design and investigate the feasibility, acceptability and safety of a digitally supported exercise maintenance intervention to Falls Management Exercise (FaME) programme service-users.

STUDY OBJECTIVES:

1. Co-design a digitally supported exercise maintenance intervention with a Community of Practice Group (COPG) and Patient and Public Involvement (PPI) group.
2. Investigate the acceptability of the digitally supported exercise maintenance intervention to FaME programme service-users.
3. Assess the feasibility of the research methods and key parameters needed to conduct future clinical trials.

STUDY DESIGN: The project will be conducted in two separate phases as interdependency exists between the research objectives:

* Phase 1. Intervention Development & Acceptability Study
* Phase 2. Feasibility Study.

METHODS:

Phase 1. Intervention development and Acceptability Study

Intervention Development will be informed by the Normalisation Process Theory and Theoretical Framework of Acceptability[1, 2]. In consultations, the investigators will work with a group of diverse PPI members and key stakeholders to define a digitally supported exercise maintenance intervention and procedures. Digital intervention components may include self-monitoring physical activity (PA) via wearables, digital peer support and home exercise delivered via an evidence-based Falls Prevention App (KOKU App).

To explore early intervention acceptability, n=10 FaME class users will be invited to test the exercise maintenance intervention for 1 month. Intervention acceptability feedback will be collected via technology acceptance questionnaires[4, 5], analysed and triangulated into a report.

After initial testing, the research participants will be invited to attend a COPG workshop, containing researchers, PPI members and service providers, to provide further qualitative feedback regarding the interventions acceptability. During the workshop, the collective group will use the participants feedback and the information in the report to optimise the intervention for progression into phase 2. Workshops will be audio-recorded, transcribed, and analysed thematically.

Phase 2. Feasibility Study:

A mixed methods single-arm multi-site feasibility study will be conducted to investigate the feasibility, acceptability and safety of the exercise maintenance intervention (optimised in phase 1) and the feasibility of the research methods.

The investigators will recruit and deliver the exercise maintenance intervention for up to 6 months in 30 FaME class attendees.

Feasibility data will be collected and measured over 6 months via:

* Recruitment and retention rates.
* Feasibility of collecting self-reported quality of life, falls incidence, and confidence data via the Falls Prevention App
* Adverse event data
* Intervention adherence will be ascertained via; i) frequency and duration of technology use and exercise progressions, ii) Weekly minutes of MVPA and strength and balance exercise minutes

A priori progression criteria will be set on feasibility outcomes to determine future progression to a larger-scale clinical trial. The progression criteria for a full-scale trial will be as follows: ≥70% of targeted number of participants are recruited within a 6-month window; ≥50% of recruited participants complete the study and provide outcome data at follow up; evidence that participants have maintained an improvement in falls risk factors; <10% of any serious adverse effects deemed to be due to the intervention.

Intervention acceptability will be qualitatively examined via semi-structured interviews with up to n=20 participants. Semi-structured interviews will be conducted by a researcher in the participants preferred venue or online. Interviews will be audio recorded, transcribed, and handled using NVIVO10-software. Two researchers will code the transcripts via framework analysis.

Participant data is routinely collected by the HealthWorks Charity for service purposes. Under information sharing agreements, the following routine data will be shared with the researchers: Age, gender, ethnicity, postcode/IMD, height, body weight, medical history, medication, falls history, functional ability (i.e. 30-s chair stand, Timed-Up-and-Go), balance measures (i.e. four-stage balance test).

Routine data will be collected at three time-points (T1-before FaME, T2-after FaME, T3-after the maintenance intervention) and will be analysed and reported via descriptive statistics.

SAMPLE & SETTING: The investigators are working in collaboration with the HealthWorks Charity that delivers FaME classes to people living in deprived areas of Newcastle Upon Tyne (England). To ensure people experiencing health inequalities are represented in the study, the investigators will recruit a sample of older adults from four HealthWorks Charity hubs and deliver the intervention in these venues.

ELIGIBILITY:
Eligibility criteria:

* Community dwelling older adults, aged over 60 years old.
* Enrolled on a Healthworks FaME programme in the Northeast region of England.
* Able to provide informed written consent.

Exclusion criteria:

* Unable to independently walk 5 metres without a walking aid.
* Advised by a medic not to undertake exercise.
* Has a medical, cognitive, or physical condition that prevents safe engagement with digital technology or unsupervised exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Seniors Technology Acceptance questionnaire (STAM) (phase 1) | after 1 month of using the KESS intervention
  Acceptability feedback on the digital health components will be collected via the Seniors Technology Acceptance questionnaire. The questionnaire contains 14 questions and statements and asks the respondent to rate their response using a 1 to 10 sliding scale (i.e. 1=strongly disagree- 10= strongly agree).
Health Intervention Acceptability Questionnaire (phase 1) | after 1 month of using the KESS intervention
  KESS intervention acceptability feedback will be collected via Health Intervention Acceptability Questionnaire. The questionnaire contains 14 questions and statements and asks respondents to rate their responses using a 1 to 5 sliding scale (i.e. 1= completely unacceptable - 5 = completely acceptable).
Physical Activity Scale for the Elderly questionnaire (PASE) | after 6 month of using the KESS intervention
  Intervention adherence will be ascertained via weekly minutes of moderate to vigorous physical activity and strength and balance exercise. The PASE questionnaire asks respondentss to provide information on the amount of physical activity they have performed for leisure, household chores and work / occupational tasks in the past 7 days.

SECONDARY OUTCOMES:
Frequency and duration of KOKU App use (Phase 2) | after 6 month of using the KESS intervention
  Intervention adherence will be ascertained via the frequency (no of times per week) and duration (weekly number of minutes) of technology use the is collected via KOKU App metrics.
Recruitment rates (phase 2) | after 6 month
  Recruitment rates will be recorded as the number of participants invited and the percentage consenting to enter the feasibility study.
Retention rates (phase 2) | during and after 6 month of using the KESS intervention
  Retention rates will be calculated as the percentage of class participants providing follow up data post intervention.
Adverse event data (Phase 2) | during the 6 month intervention period
  Adverse event data will be collected by the research team monthly (via email and telephone) and assessed by the Principal Investigator and Clinical Leads for causality to determine if events are related to the interventions receipt.
Fear of falling questionnaire completion (Phase 2) | Questionnaire completion will be measured at baseline and post intervention (6-months).
  Feasibility of self-reported fear of falling data via the KOKU App will be determined by the number and percentage of participants completing the inbuilt questionnaires on fear of falling
Falls incidence questionnaire completion (Phase 2) | Questionnaire completion will be measured at baseline and post intervention (6-months).
  Feasibility of collecting self-reported falls incidence data via the KOKU App will be determined by the number and percentage of participants completing the inbuilt questionnaires on falls incidence.
Quality of life questionnaire completion (Phase 2) | Questionnaire completion will be measured at baseline and post intervention (6-months).
  Feasibility of collecting self-reported quality of life data via the KOKU App will be determined by the number and percentage of participants completing the inbuilt questionnaires on quality of life.
Semi-structured interviews regarding KESS Acceptability | after the 6 month intervention period.
  Intervention acceptability will be qualitatively examined via semi-structured interviews with up to n=20 participants. Interview Schedules will be informed by the Theoretical Framework of Acceptability and Seniors Technology Acceptance Model.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthWorks: The Health Resource Centre, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No